CLINICAL TRIAL: NCT05418920
Title: Comparing the Efficacy of Double-flap Technique Versus Single-flap Technique After Proximal Gastrectomy: a Multicentre Randomized Controlled Trial
Brief Title: Clinical Trial of Reconstruction After Proximal Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncogastroenterology Committee of Chinese (Other)
Collaborators: Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); General Hospital of Ningxia Medical University (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: single-flap technique
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Esophagitis, Reflux
Keywords: left open single-flap technique, proximal gastrectomy
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the trial group (left-opening single-flap group) (Experimental): left-opening single-flap group
  Interventions: Procedure: left-opening single-flap technique
- the control group (double-flap group) (Active Comparator): double-flap group
  Interventions: Procedure: double-flap group technique

INTERVENTIONS:
Procedure: left-opening single-flap technique — left-opening single-flap technique
  Arms: the trial group (left-opening single-flap group)
Procedure: double-flap group technique — double-flap group technique
  Arms: the control group (double-flap group)

SUMMARY:
1) To explore a simple, safe, post-proximal gastrectomy reconstruction method with good absorption and digestive function in order to improve patients' postoperative quality of life; 2) To fill the gap in the comparison of clinical efficacy between left-open single-flap technique and double-flap technique in this specialized field in China; 3) To utilize the experience and foundation of gastrointestinal surgery in the treatment of gastric cancer and integrate the advantageous resources in China; 4) To establish a large-sample, multicenter randomized clinical study in order to promote the establishment and improvement of relevant norms of gastrointestinal reconstruction

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common cancer worldwide and the third leading cause of cancer-related deaths each year. Although the incidence of gastric cancer has decreased worldwide compared to the past, the incidence of esophagogastric junction cancer and upper 1/3 gastric cancer is gradually increasing. Currently, the main treatment for esophagogastric junction cancer and upper gastric cancer is surgery. However, there is no clinical consensus on the choice of surgical approach for these patients. Compared with total gastrectomy, proximal gastrectomy can preserve the physiological function of the stomach and has great advantages in nutrient absorption, thus it has been widely accepted in Asian countries.

However, the risk of developing reflux esophagitis after proximal gastrectomy is high, which seriously affects patients' postoperative quality of life. In order to reduce the occurrence of postoperative complications, clinicians continue to improve the methods of GI reconstruction. Currently, the common methods of GI reconstruction after proximal gastrectomy include esophagogastrostomy (EG), jejunal intubation (JI), jejunal pouch intubation (JPI), and dual-tract reconstruction (DTR). However, the choice of the optimal reconstruction method after proximal gastrectomy remains controversial, and there is no standard approach to GI reconstruction. In 2016, Kuroda et al. reported a new surgical approach with a double-flap technique after proximal gastrectomy and showed satisfactory short-term outcomes compared with conventional esophagogastric anastomosis. At the 1-year postoperative follow-up, no reflux esophagitis was detected in all patients. At the same time, the rate of anastomotic stenosis was noteworthy.

This study will be the first attempt at a left-open single-flap technique, which was modified from the double-flap technique. The short-term outcome was satisfactory in all patients. This study will establish a large sample, multicenter randomized clinical study. By exploring a simple, safe, good absorption and digestive function method of post-proximal gastrectomy reconstruction to improve patients' postoperative quality of life and fill the gap in the comparison of clinical efficacy between left-open single-flap technique and double-flap technique in this specialized field. This will promote the establishment and improvement of the specifications related to gastrointestinal reconstruction.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 18-80 years, regardless of gender;
2. Siewert III of the esophagogastric junction adenocarcinoma: Stage Ⅰ(cT1-2N0M0) or adenocarcinoma of the upper part of the stomach： Stage Ⅰ(cT1-2N0M0), Stage II( cT1-2N1-3M0 / cT3-4N0M0), Stage III(cT3-4aN1-3M0); patients who are suitable for surgery according to the 8th AJCC clinical staging of gastric cancer;
3. Primary lesion diagnosed by preoperative endoscopic end pathology: tumor diameter <4 cm and located in the upper part of the stomach (including the esophagogastric junction), histologically confirmed adenocarcinoma;
4. Preoperative ASA score: I, II, or III;
5. Preoperative Karnofsky physical status score: ≥ 70%; or preoperative ECOG physical status score: ≤ 2;
6. No distant metastases (confirmed by preoperative chest X-ray, abdominal ultrasound, and upper abdominal CT); no peritoneal implant metastases (confirmed by laparoscopic exploration surgery);
7. R0 surgical outcome is expected to be obtained with radical gastrectomy of D2 proximal gastric cancer;
8. Patients and their families voluntarily participate in this study and sign the informed consent form after understanding the study content.

Exclusion Criteria

1. Patients received any preoperative treatment, such as chemotherapy, radiotherapy, targeted therapy or immunotherapy; preoperative neoadjuvant chemotherapy recipients;
2. Patients with clinical stage exceeding Siewert III of the esophagogastric junction adenocarcinoma: Stage Ⅰ(cT1-2N0M0) or more than adenocarcinoma of the upper part of the stomach: Stage Ⅰ(cT1-2N0M0), Stage II(cT1-2N1-3M0/cT3-4N0M0), Stage III(cT3-4aN1-3M0);
3. Patients with acute infections, especially biliary tract infections;
4. Patients with complications of gastric cancer (bleeding, perforation, obstruction) requiring emergency surgery;
5. Patients with uncorrectable coagulation dysfunction;
6. Patients with vital organ failure, such as heart, lung, liver, brain, kidney, etc.
7. Severe central nervous system disease, mental disorders, or impaired consciousness;
8. Pregnant or lactating women;
9. Patients with distant metastases;
10. Patients with a primary tumor at another site diagnosed within the past 5 years;
11. Preoperative ASA score: ≥ IV;
12. Preoperative ECOG physical status score: ≥ 2;
13. History of continuous systemic corticosteroid therapy within the past 1 month;
14. History of unstable angina, myocardial infarction, cerebral infarction, or cerebral hemorrhage within the past 6 months;
15. Patients with concurrent surgical treatment of other diseases;
16. Patients with immunodeficiency, immunosuppression, or autoimmune diseases (organ transplant requiring immunosuppressive therapy within the past 5 years, allogeneic bone marrow transplant patients, taking immunosuppressive drugs, etc.);
17. Patients with concurrent participation in other clinical studies;
18. Patients refusing to sign an informed consent form to participate in this study;
19. Preoperative imaging: regional fusion of enlarged lymph nodes (maximal diameter > 3 cm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of reflux esophagitis | 12 months
  Incidence of reflux esophagitis

SECONDARY OUTCOMES:
Overall postoperative complication rate | 30 days
  Overall postoperative complication rate
Incidence of anastomotic fistula | 30 days
  Incidence of anastomotic fistula
Operation time | intraoperative
  Operation time
Bleeding loss volume | intraoperative
  Bleeding loss volume
incidence of anastomotic stricture | 30 days
  incidence of anastomotic stricture
Incidence of reflux esophagitis | 6 days
  Incidence of reflux esophagitis

CONTACTS AND LOCATIONS:
Overall Officials: Nan Wang, MD, Study Chair — Tang-Du Hospital; Chao Zhang, MD, Study Chair — Henan Provincial People's Hospital; Lei Wang, MD, Study Chair — General Hospital of Ningxia Medical University; Renwei Chang, MD, Study Chair — The First Affiliated Hospital of Shanxi Medical University; Junjun She, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

REFERENCES:
- [Derived] Yang QC, Wang WD, Mo ZC, Yue C, Zhou HK, Gao RQ, Yu J, Dong DH, Liu JQ, Wei JP, Yang XS, Ji G, Li XH. Study protocol for comparing the efficacy of left-open single-flap technique versus double-flap technique after proximal gastrectomy: A multicenter randomized controlled trial. Front Oncol. 2022 Nov 17;12:973810. doi: 10.3389/fonc.2022.973810. eCollection 2022. PMID 36465382